CLINICAL TRIAL: NCT02545270
Title: Validation of a Subjective Rating Scale for Assessment of the Surgical Workspace in Laparoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Roar Medici, Research Assistant, MD., Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Vallap01
Record Dates: First submitted 2015-08-06; First posted 2015-09-09 (Estimated); Results first posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-03

CONDITIONS: Hernia, Inguinal
Keywords: Surgery, Laparoscopic; surgical rating scale
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1: 12-9-6 mmHg (Experimental): Elective laparoscopic inguinal hernia procedures will be used to make three video-recordings (lasting 20-30 seconds) under different levels of pneumoperitoneum (12-9-6 mmHg) during desufflation after surgery is completed.
  Interventions: Procedure: Level of pneumoperitoneum 12-9-6 mmHg
- Group 2: 11-8-5 mmHg (Experimental): Elective laparoscopic inguinal hernia procedures will be used to make three video-recordings (lasting 20-30 seconds) under different levels of pneumoperitoneum (11-8-5 mmHg) during desufflation after surgery is completed.
  Interventions: Procedure: Level of pneumoperitoneum 11-8-5 mmHg
- Group 3: 10-7-4 mmHg (Experimental): Elective laparoscopic inguinal hernia procedures will be used to make three video-recordings (lasting 20-30 seconds) under different levels of pneumoperitoneum (10-7-4 mmHg) during desufflation after surgery is completed.
  Interventions: Procedure: Level of pneumoperitoneum 10-7-4 mmHg

INTERVENTIONS:
Procedure: Level of pneumoperitoneum 12-9-6 mmHg — Elective laparoscopic inguinal hernia procedures will be used to make video-recordings under 3 different levels of pneumoperitoneum (12-9-6 mmHg) during desufflation.
  Arms: Group 1: 12-9-6 mmHg
Procedure: Level of pneumoperitoneum 11-8-5 mmHg — Elective laparoscopic inguinal hernia procedures will be used to make video-recordings under 3 different levels of pneumoperitoneum (11-8-5 mmHg) during desufflation.
  Arms: Group 2: 11-8-5 mmHg
Procedure: Level of pneumoperitoneum 10-7-4 mmHg — Elective laparoscopic inguinal hernia procedures will be used to make video-recordings under 3 different levels of pneumoperitoneum (10-7-4 mmHg) during desufflation.
  Arms: Group 3: 10-7-4 mmHg

SUMMARY:
It is of great importance to obtain optimal surgical conditions for the surgeon in order to increase patient safety. The effect of different interventions on surgical conditions has been assessed by various surgeon-assessed rating scales. A 5-point surgical rating scale has previously been tested in a proof-of-concept trial - but not validated - during radical retropubic prostatectomy by asking different surgeons to evaluate the surgical workspace using video sequences.

In an ongoing study (The Hernia Study, Trial registration NCT02247466) performed by investigators group, investigators are using a 5-point scale to rate the surgical workspace during laparoscopic ventral herniotomy with or without neuromuscular blockade. This scale is based on previously used scales by already published studies and has a description connected to each point. To the authors' knowledge the scale has never been validated in a laparoscopic setting, where the intra-abdominal pressure during pneumoperitoneum can have a great influence on visualization. In fact, to investigators knowledge, no validated surgeon-assessed rating scale regarding the surgical workspace during laparoscopic surgery does exists.

Purpose:

Primary aim:

To validate a 5-point rating scale by investigating the inter-rater agreement of evaluations of the surgical workspace at different intra-abdominal pressures. Using intra-abdominal video recordings.

Secondary aims:

To validate a 10-point rating scale by investigating the inter-rater agreement of evaluations of the surgical workspace at different intra-abdominal pressures.

To test the agreement between the two rating scales. To assess which of the two rating scales has the highest inter-rater agreement To assess the intra-rater agreement of both rating scales.

Hypothesis:

Investigators hypothesize that the 5-point rating scale has an intra-class correlation coefficient (ICC) > 0.6., validated by video-sequences obtained during laparoscopic surgery.

DETAILED DESCRIPTION:
Scales:

The 5-point scale used to assess the surgical workspace during laparoscopic herniotomy:

1. (Extremely poor conditions) Unable to complete surgery without interventions*
2. (Poor conditions) Several minor adjustments needed to complete surgery. (ie. changes in patient positioning, surgeon position)
3. (Acceptable conditions) After few minor adjustments surgery can be completed.
4. (Good conditions) Surgical workspace is good, but there is some interference, but no need for adjustments.
5. (Optimal conditions) Surgical workspace is optimal and procedure can be completed without any interference.

   * Interventions are defined as change in depth of neuromuscular blockade and/or pneumoperitoneum.

The 10-point scale used to assess the surgical workspace during laparoscopic herniotomy is a Visual Analog Scale, where the surgeon specify their rating of the surgical workspace by indicating a position along a continuous line between two end-points

Video recordings:

Elective laparoscopic inguinal hernia procedures will be used to make video-recordings under different levels of pneumoperitoneum during desufflation after surgery is completed.

Each video-sequence will last 20-30 seconds and. three video-sequences during different levels of pneumoperitoneum will be made from each patient. The patients are randomized to one of three groups regarding level of pneumoperitoneum during the three video-recordings. Group 1: 12-9-6 mmHg, 2: 11-8-5, 3: 10-7-4 mmHg. Three video-sequences during different levels of pneumoperitoneum (according to group allocation) will be made from each patient.

We will record 5 pilot video-sequences and have them evaluated by two experienced surgeons in order to design a standard setup for filming the surgical workspace.

From the 30 recorded video-sequences investigators will choose the 24 video-sequences best illustrating different levels of surgical workspace.

The video-sequences will be embedded in an internet form, and each sequence is followed by a question about the rating of that particular surgical workspace.

Each surgeon will be presented to the 24 sequences in a randomly selected recordings of different patients. After each recording the surgeon will evaluate the surgical work space on one of the two rating scales. After rating all recordings, using one scale, the recordings will repeat in a random order and the second scale should be used. When doing the assessment the surgeon should imagine that he/she is about to do a laparoscopic inguinal herniotomy, and the evaluation/rating is based on this situation.

The surgeons are not allowed to discuss their ratings with each other during the study.

To observe intra-rater agreement the surgeon will assess the same sequence at least twice using the same rating scale. Therefore the surgeons will see all recordings four times during the study.

Sample size requirements are calculated by estimating the width of the confidence interval(CI) as described by Shoukri et all. An ICC of 0.8 with a 95% CI of [0.6-1.0] can be achieved with 8 surgeons assessing 24 recordings. To ensure sufficient variation in the recordings investigators will include a total of 10 patients and make three recordings from each.

Sample size requirements are calculated by estimating the width of the confidence interval(CI) as described by Shoukri et all. An ICC of 0.8 with a 95% CI of [0.6-1.0] can be achieved with 8 surgeons assessing 24 recordings. To ensure sufficient variation in the recordings we will include a total of 10 patients and make three recordings from each. Investigators assume that the 24 recordings can be seen as 24 independent subjects.

Both the inter-rater agreement and the intra-rater agreement will be calculated using Kappa and intraclass correlation statistics. with statistical software6. The model for ICC will be a two-way random, single measures, absolute agreement, ( ICC(2,1) ) Calculated using SPSS (ver 22.0).

The agreement between the two rating scales will be tested with regression analysis using Spearman correlation coefficient.

To assess which of the two rating scales that has the highest inter-rater agreement the two scales corresponding ICC with confidence intervals will be compared.

Investigator and co-authors will be responsible for analyzing the study data with assistance from Statistician located at Herlev Hospital.

Investigators will include 8 surgeons (Specialist level of training and proficient in laparoscopic inguinal surgery).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* Elective laparoscopic inguinal herniotomy.
* Can read and understand Danish

Exclusion Criteria:

* Technical difficulties making video recording impossible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-03; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roar Medici, MD, Principal Investigator — Herlev Hospital University of Copenhagen
Locations (2):
- Denmark (2):
  - Gentofte Hospital, Hellerup, Capital Region
  - Herlev Hospital, Copenhagen

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1: 12-9-6 mmHg | Group 2: 11-8-5 mmHg | Group 3: 10-7-4 mmHg
Started | 6 | 5 | 5
Completed | 6 | 4 | 3
Not Completed | 0 | 1 | 2
Not completed — technical difficulties | 0 | 1 | 0
Not completed — Videos being too similar to other | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Demographics for patients whose videos were embedded in the questionnaire.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: 12-9-6 mmHg | Group 2: 11-8-5 mmHg | Group 3: 10-7-4 mmHg | Total
Number analyzed (Participants) | 6 | 5 | 5 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 3 | 3 | 6
  >=65 years | 6 | 2 | 2 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1
  Male | 5 | 5 | 5 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 6 | 5 | 5 | 16
ASA score [Count of Participants; unit: Participants] — American Society of Anaesthesiologists (ASA) physical status classification system. Ranged from 1-5; 1 is best
  Participants
    ASA 1 | 4 | 3 | 3 | 10
    ASA 2 | 2 | 2 | 2 | 6
Neuromuscular blockade used [Count of Participants; unit: Participants]
  Neurosmuscular blockade used | 3 | 3 | 0 | 6
  Neurosmuscular blockade NOT used | 3 | 2 | 5 | 10
Type of anesthesia [Count of Participants; unit: Participants] — Total intravenous anesthesia (TIVA) or not TIVA
  Participants
    TIVA | 5 | 5 | 5 | 15
    Not TIVA | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Inter-rater Agreement, 5-point Scale
Description: To validate a 5-point rating scale by investigating the inter-rater agreement of evaluations of the surgical workspace at different intra-abdominal pressures.
  The 5-point surgical rating scale is categorical, with following descriptions: 1 (Extremely poor conditions) Unable to complete surgery without interventions 2 (Poor conditions) Several minor adjustments needed to complete surgery. (e.g. changes in patient body position, surgeon position) 3 (Acceptable conditions) After few minor adjustments surgery can be completed. 4 (Good conditions) Surgical workspace is good, but there is some interference, but no need for adjustments.
  5 (Optimal conditions) Surgical workspace is optimal and procedure can be completed without any interference.
  Using intra-abdominal video recordings. The inter-rater agreement will be calculated using intraclass correlation statistics with statistical software.
Time Frame: 60 min
Population: The 24 videos recorded from 13 participants.
Measure: Number (95% Confidence Interval); unit: ICC
Units Other Than Participants: Videos
Groups:
- Surgeons Assessing Video Sequences: 7 experienced surgeons recruited: Specialist level of training Performed >200 laparoscopic cholecystectomies
Arm/Group | Surgeons Assessing Video Sequences
Number analyzed (Participants) | 13
Number analyzed (Videos) | 24
ICC | 0.57 [0.45 to 0.69]

2. Secondary Outcome: Inter-rater Agreement, 10-point Scale
Description: To validate a 10-point rating scale by investigating the inter-rater agreement of evaluations of the surgical workspace at different intra-abdominal pressures. The inter-rater agreement will be calculated using intraclass correlation statistics with statistical software.
  The 10-point rating scale was a discrete numerical scale with 1 being worst possible surgical workspace and 10 being best possible.
Time Frame: 60 min
Population: The 24 videos recorded from 13 participants.
Measure: Number (95% Confidence Interval); unit: ICC
Units Other Than Participants: Videos
Arm/Group | Surgeons Assessing Video Sequences
Number analyzed (Participants) | 13
Number analyzed (Videos) | 24
ICC | 0.54 [0.39 to 0.58]

3. Secondary Outcome: Agreement Between the Two Rating Scales Will be Tested With Regression Analysis Using Spearman Correlation Coefficient
Description: The agreement between the two rating scales 5-point categorical and 10-point numerical will be tested with regression analysis using Spearman correlation coefficient
Time Frame: 60 min
Population: Agreement between the two rating scales ( 5-poit categorical and 10-point numerical) used to assess the 24 videos recorded from 13 participants.
Measure: Number (95% Confidence Interval); unit: Spearman correlation coefficient
Units Other Than Participants: Scales
Groups:
- Strength of the Relationship Between the Two Scales: A regression analysis using Spearman's correlation coefficient was calculated to assess the strength of the relationship between the two scales.
Arm/Group | Strength of the Relationship Between the Two Scales
Number analyzed (Participants) | 13
Number analyzed (Scales) | 2
Spearman correlation coefficient | 0.79 [0.56 to 0.90]

4. Secondary Outcome: Intra-rater Agreement of Both Rating Scales.
Description: To assess the intra-rater agreement of both rating scales, 10-point numerical and 5-point categorical scale.
  The intra-rater agreement will be calculated using intraclass correlation statistics.
Time Frame: 60 min
Population: Intra-rater agreement of both scales ( 5-poit categorical and 10-point numerical) used to assess the 24 videos recorded from 13 participants.
Measure: Number (95% Confidence Interval); unit: ICC
Groups:
- Surgeons Assessing Video Sequences 5-point Scale; Surgeons Assessing Video Sequences 10-point Scale: 7 experienced surgeons recruited: Specialist level of training Performed >200 laparoscopic cholecystectomies
Arm/Group | Surgeons Assessing Video Sequences 5-point Scale | Surgeons Assessing Video Sequences 10-point Scale
Number analyzed (Participants) | 13 | 13
ICC | 0.78 [0.71 to 0.84] | 0.84 [0.8 to 0.88]

ADVERSE EVENTS:
Time Frame: Through video-recording completion, an average of half an hour
Arm/Group | Group 1: 12-9-6 mmHg | Group 2: 11-8-5 mmHg | Group 3: 10-7-4 mmHg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/6 | 0/4 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No